CLINICAL TRIAL: NCT00439452
Title: Telemedicine-Based Collaborative Care to Reduce Rural Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 61251
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine-Based Collaborative Care (Active Comparator): Telemedicine-Based Collaborative Care - Off-site depression care team (telephone nurse care manager, telephone pharmacist, tele-psychologist and tele-psychiatrist) works collaboratively with on-site primary care providers. Telephone nurse care manager activities include promoting patient activation and self management, assessing symptoms and comorbidities, and monitoring adherence, side-effects and treatment response. Telephone pharmacist activities include documenting medication histories and conducting medication management. Tele-psychologist activities include providing cognitive behavioral therapy via interactive video. Tele-psychiatrist activities include conducting patient consultation via interactive video.
  Interventions: Other: Telemedicine-Based Collaborative Care
- Practice Based Collaborative Care (Active Comparator): One-site nurse care manager works collaboratively with on-site primary care providers. Nurse care manager activities include promoting patient activation and self management, assessing symptoms and comorbidities, and monitoring adherence, side-effects and treatment response.
  Interventions: Other: Practice Based Collaborative Care

INTERVENTIONS:
Other: Telemedicine-Based Collaborative Care — Off-site depression care team (telephone nurse care manager, telephone pharmacist, tele-psychologist and tele-psychiatrist) works collaboratively with on-site primary care providers. Telephone nurse care manager activities include promoting patient activation and self management, assessing symptoms and comorbidities, and monitoring adherence, side-effects and treatment response. Telephone pharmacist activities include documenting medication histories and conducting medication management. Tele-psychologist activities include providing cognitive behavioral therapy via interactive video. Tele-psychiatrist activities include conducting patient consultation via interactive video.
  Arms: Telemedicine-Based Collaborative Care
Other: Practice Based Collaborative Care — One-site nurse care manager works collaboratively with on-site primary care providers. Nurse care manager activities include promoting patient activation and self management, assessing symptoms and comorbidities, and monitoring adherence, side-effects and treatment response.
  Arms: Practice Based Collaborative Care

SUMMARY:
Across the country, Community Health Centers are participating in the Health Disparities Collaboratives sponsored by the Health Services Resources and Services Administration (HRSA). The Health Disparities Collaboratives integrate three complementary conceptual frameworks: 1) the Institute for Healthcare Improvement's (IHI) Breakthrough Series Model; 2) the Improvement Model (i.e., Plan-Do-Study-Act cycles); and 3) Wagner's Chronic Care Model. The Chronic Care model uses patient self-management, delivery system re-design, decision support, and clinical information systems to maximize the effectiveness of interactions between prepared proactive care teams and informed activated patients with chronic illnesses such as diabetes, asthma, and depression. The Chronic Care model for depression, also known as Collaborative Care, involves primary care providers working with a depression care team comprising non-physicians (e.g., nurses, pharmacists) and mental health specialists (e.g., psychiatrists). Practice-based collaborative care involves primary care providers working with an on-site depression care team. In contrast, telemedicine-based collaborative care involves primary care providers working with an off-site depression care team using telemedicine technologies. The purpose of this research project is to compare the effectiveness and cost effectiveness of practice-based and telemedicine-based collaborative care in Community Health Centers (without on-site mental health specialists) implementing the Health Disparities Collaborative for depression.

DETAILED DESCRIPTION:
An experimental study design and an intent-to-treat analysis will be used to determine the effectiveness and cost-effectiveness of telemedicine-based collaborative care relative to practice-based collaborative care. The research setting will be six Community Health Centers located in medically underserved areas of Arkansas which serve rural, low income and minority populations. Potentially eligible patients will be identified through screening by Community Health Centers clinic staff or primary care provider referrals. Patients eligible for the study will be consented and randomized to receive either telemedicine-based or practice-based collaborative care, and followed for 18 months to assess processes and outcomes. On-site clinical staff will screen patients for depression over an 18 month period and refer all patients with clinically significant depression (PHQ9≥10) to the study.

Two types of health care professionals will be involved in the practice-based collaborative care model: 1) primary care providers (MD and RNP); and 2) a depression care manager (LPN or Social Worker). The on-site care managers will provide care management activities by phone or face-to-face.

Five types of health care professionals will be involved in the telemedicine-based collaborative care model: 1) primary care providers (MD and RNP); 2) a depression nurse care manager (RN); 3) clinical pharmacist (PharmD); 4) tele-psychologist (PhD); and 5) a tele-psychiatrist (MD). The primary care providers will be located at the Community Health Centers. The off-site depression care team will be located at the clinics of the University of Arkansas for Medical Sciences, Department of Psychiatry. The on-site primary care providers will prescribe medications and schedule all appointments. The off-site nurse care manager will conduct all care management activities by telephone. The off-site clinical pharmacist will conduct medication histories and provide medication management by telephone. The off-site tele-psychologist will conduct evidence-based psychotherapy (cognitive behavioral therapy) via interactive video. The off-site tele-psychiatrist will conduct interactive-video consultations, train and supervise the depression care team, and conduct provider education.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Significant Depression

Exclusion Criteria:

* Sub-threshold Depression,
* Non-english speaking,
* Patients not having telephone access,
* Bereaved,
* Suicidal,
* Currently being treated by a mental health specialist,
* Bipolar disorder,
* Psychotic disorders,
* Drug or alcohol dependence,
* Cognitively impaired,
* Terminal illness,
* Having a court appointed guardian, or
* Pregnant (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare processes and outcomes between CHC patients receiving practice-based collaborative care to CHC patients receiving telemedicine-based collaborative care (OUTREACH intervention). | 6, 12, 18 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: John C Fortney, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Mittal D, Chekuri L, Lu L, Fortney JC. Demographic, Economic, and Clinical Correlates of Depression Treatment Response in an Underserved Primary Care Population. J Clin Psychiatry. 2014 Aug 26;75(8):848-854. doi: 10.4088/JCP.13m08954. PMID 29676557
- [Derived] Grubbs KM, Fortney JC, Pyne J, Mittal D, Ray J, Hudson TJ. A Comparison of Collaborative Care Outcomes in Two Health Care Systems: VA Clinics and Federally Qualified Health Centers. Psychiatr Serv. 2018 Apr 1;69(4):431-437. doi: 10.1176/appi.ps.201700067. Epub 2018 Jan 16. PMID 29334874
- [Derived] Pyne JM, Fortney JC, Mouden S, Lu L, Hudson TJ, Mittal D. Cost-effectiveness of on-site versus off-site collaborative care for depression in rural FQHCs. Psychiatr Serv. 2015 May 1;66(5):491-9. doi: 10.1176/appi.ps.201400186. Epub 2015 Feb 17. PMID 25686811
- [Derived] Fortney JC, Pyne JM, Mouden SB, Mittal D, Hudson TJ, Schroeder GW, Williams DK, Bynum CA, Mattox R, Rost KM. Practice-based versus telemedicine-based collaborative care for depression in rural federally qualified health centers: a pragmatic randomized comparative effectiveness trial. Am J Psychiatry. 2013 Apr;170(4):414-25. doi: 10.1176/appi.ajp.2012.12050696. PMID 23429924
- [Derived] Deen TL, Fortney JC, Schroeder G. Patient acceptance of and initiation and engagement in telepsychotherapy in primary care. Psychiatr Serv. 2013 Apr 1;64(4):380-4. doi: 10.1176/appi.ps.201200198. PMID 23370530